CLINICAL TRIAL: NCT03869372
Title: Cerebral Cortical Influences on Autonomic Function
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Levinthal (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, David Levinthal, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY19010027; 5K08DK101756-05 (NIH)
Record Dates: First submitted 2019-02-19; First posted 2019-03-11 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Healthy Subjects; Functional Dyspepsia; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Subjects will act as their own controls: The investigators will assess measures of autonomic function at baseline and in response to various modes of TMS exposure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study subjects (Experimental): At the baseline session, measures of autonomic activity (electrogastrogram - EGG, electrocardiogram - ECG, cardiac impedance - CI) will be monitored from about 15 minutes before up to 1 hour after consumption of a test meal, water or a nutrient drink. In addition, motor-evoked potentials (MEPs) elicited with single pulse transcranial magnetic stimulation will be assessed before and after the meal or drink.
  In subsequent sessions, repetitive transcranial magnetic stimulation (rTMS) is applied before the meal or drink. Based on responses to symptom surveys (IBS-SSS and PAGI-SYM), study subjects will be characterized as healthy or as having functional dyspepsia and/or IBS.
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS — In subsequent sessions, the same measures of autonomic activity and MEPs will be monitored but different patterns of repetitive TMS (rTMS) will be applied to motor cortex or other areas before the test meal, water or nutrient drink is consumed.

SUMMARY:
This is an exploratory neurophysiological study that will determine the impact of non-invasive brain stimulation on autonomic regulation, with a focus on gastrointestinal function. These studies should provide a basis for future brain-based neurotherapeutic strategies in patients with functional GI disorders.

DETAILED DESCRIPTION:
The overall goal of this study is to determine the impact of non-invasive brain stimulation on autonomic function in human subjects without functional gastrointestinal disorders and in subjects with Irritable Bowel Syndrome (IBS) or Functional Dyspepsia (FD).

Aim 1: Determine whether repetitive transcranial magnetic stimulation (rTMS) of specific cortical areas alters physiologic measures of gastrointestinal and cardiac function.

The investigators will use rTMS to transiently induce changes in neural excitability within specific cortical regions identified as being linked to autonomic regulation. Based on preliminary neuroanatomical data, one of the leading candidate cortical areas associated with sympathetic regulation lies within the trunk representation of the primary motor cortex. Thus, the investigators first plan on targeting this region of the primary motor cortex with rTMS and assess the effect of various parameters of rTMS on gastrointestinal and cardiac function in healthy human subjects. The investigators will then perform additional experiments using rTMS targeted to other specific cortical sites, such as the dorsal premotor area and rostral cingulate cortex that have also been linked to autonomic control. Each of these identified cortical regions may make unique contributions to autonomic reactivity.

Aim 2: Determine whether patients with functional gastrointestinal disorders demonstrate altered physiological reactivity to targeted rTMS.

The investigators will use the optimal parameters of rTMS and regions of interest determined in Aim 1 to assess the gastrointestinal and cardiac reactivity in participants with functional dyspepsia (FD) and/or irritable bowel syndrome (IBS). These physiological responses will be correlated with assessments of disease severity, mood, and quality of life.

--This study description has been revised since its original posting. Because all study procedures are performed in all subjects, regardless of being a healthy subject or one with FD and/or IBS, rather than a three arm trial, this trial should be regarded as having a single arm study design.

ELIGIBILITY:
Inclusion Criteria:

* Adults between age 21 and 60
* Participants without gastrointestinal symptoms (Healthy Subjects)
* Participants with gastrointestinal symptoms compatible with functional dyspepsia (FD) and or irritable bowel syndrome (IBS)

Exclusion Criteria:

* history of myocardial infarction, supplemental oxygen requirement, or diabetes
* history of chronic gastrointestinal symptoms (for healthy subjects only)
* history of gastric surgery
* psychosis or altered cognitive status
* history of head injury, metal in the skull, stroke, or a history of seizures
* implantable devices, such as a pacemaker or nerve stimulator
* current use of the following medications or use of substances which are known to lower the seizure threshold: amitriptyline (Elavil), nortriptyline (Pamelor), imipramine (Tofranil), doxepin (Sinequan), clozapine (Clozaril), chlorpromazine (Thorazine), amphetamines or methamphetamine, Ecstasy, Ketamine, Angel Dust/phencyclidine (PCP), cocaine, or 3 or more alcoholic drinks per day
* pregnancy
* Body-Mass-Index (BMI) > 35

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 244 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2026-10-03 (Estimated); Study Completion 2026-10-03 (Estimated)

PRIMARY OUTCOMES:
Electrogastrogram (EGG) | EGG will be monitored for 15 minutes before and up to 1 hour after consumption of the nutrient drink or the test meal
  The EGG will be analyzed in the frequency domain using fast Fourier Transformation (FFT). The power spectrum will be divided into frequency bands (normal gastric activity (~3 cycles per minute), slower than normal (bradygastria) and faster than normal (tachygastria)). rTMS-induced shifts in the power distribution across these frequency bands after consumption of water or a nutrient drink or a test meal will be compared to water or nutrient drink or test meal without rTMS.
Volume threshold to satiety | volumes will be determined immediately after the 5 min drinking window and compared across study sessions
  rTMS-induced shift in the volume of water or nutrient drink a subject can consume within a 5 min period before reaching satiety

SECONDARY OUTCOMES:
MEP responses | before and up to 1 hour after rTMS
  rTMS-induced change in the amplitude of motor evoked potentials (MEP) elicited by single pulse TMS
Heart rate variability | before and up to 1 hour after rTMS
  rTMS-induced change in heart rate variability elicited by Valsalva maneuver or diaphragmatic breathing
Cardiac Impedance | before and up to 1 hour after rTMS
  rTMS-induced change in cardiac impedance variability

CONTACTS AND LOCATIONS:
Overall Officials: David J Levinthal, MD/PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
There is no current plan to share with specific individuals, but individual participant data and supporting information (below) that are the basis for the published results will be made available after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months after article publication and up to 5 years thereafter.
Access Criteria: Proposals to access trial data should be directed to the Principal Investigator (Dr. David Levinthal) at levinthald@upmc.edu, and if the researcher has a sound basis for the proposal, then requestors will be asked to sign a data access agreement (link to be determined).